CLINICAL TRIAL: NCT00265603
Title: Phase 1 Toxicity/Feasibility Study: Combined Modality Treatment With Transimmunization for Non-Small Cell Lung Cancer
Brief Title: Safety Study: Combined Modality Treatment for Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R04-10-009
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Arm (Experimental): The investigators plan to have approximately 16 persons participate in the study of transimmunization. Transimmunization uses a device, called a UVAR-XTS instrument, to remove a portion of blood, part of which is returned, and part of which is incubated overnight before being returned to the bloodstream the next day
  Interventions: Procedure: Extracorporeal Photochemotherapy With Transimmunization

INTERVENTIONS:
Procedure: Extracorporeal Photochemotherapy With Transimmunization — The photopheresis apparatus and procedure will be identical to that currently used. Patients will receive intravenous 8-MOP (UVADEX®) directly into the photopheresis apparatus, to yield a concentration of 50-200 ng/ml of drug. The blood will be leukapheresed to obtain a buffy coat and will then be passed through the contiguous closed circuit ultraviolet A exposure device, delivering the desired 1-2 joules/cm2 of ultraviolet A energy. In this manner 2-4 molecules of 8-MOP will be induced to bind covalently to thymines of the leukocyte DNA. At that point, the single variation from the standard treatment will be initiated. Instead of returning the patient's cells and the saline to the patient, the bag will be detached from the apparatus. KLH (depyrogenated, endotoxin-free; Calbiochem-Novabiochem Corp., San Diego, CA) will be added at a concentration of 10 g/ml to the DC-rich leukocyte culture prior to overnight culture.

SUMMARY:
The purpose of this study is to determine the safety of using a treatment called transimmunization in addition to standard therapy (radiation) in the treatment of lung cancer. Transimmunization is a treatment of the blood designed to boost the immune response against lung cancer. Transimmunization uses a device called a UVAR-XTS instrument, to remove a portion of blood, part of which is returned, and part of which is incubated overnight before being returned to the bloodstream the next day.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in both men and women in the United States. It is estimated that there are over 170,000 new cases of lung cancer in the United States and over 150,000 deaths annually. Surgical excision is currently the treatment of choice for patients with operable non-small cell lung cancer (NSCLC). However, only a minority of patients present with early stage, surgically resectable disease. Most patients present with advanced disease confined to the chest, but not surgically resectable (Stage IIIB), or metastatic disease (Stage IV). Conventional treatment for stage IIIB NSCLC is concurrent or sequential radiation therapy and chemotherapy, while standard treatment for stage IV disease is chemotherapy therapy alone, with radiation therapy for palliative adjunctive treatment. Currently, five-year survival rates for patients with Stage IIIB and IV disease, treated or untreated, is less than 15%. We propose herein a Phase I trial to assess the safety of Transimmunization as a component of combined modality treatment for stage IIIB or IV NSCLC by incorporating this immunotherapy with radiotherapy.

Extracorporeal photochemotherapy (ECP), or photopheresis, was originally introduced for the management of patients with cutaneous T cell lymphoma (CTCL). In the fifteen years since it became the first FDA approved tumor-targeting selective immunotherapy for the treatment of any cancer, it has induced partial responses in a majority of the erythrodermic CTCL patients with residual immunocompetence to whom it has been administered (in more than 150 centers, more than 250,000 times) throughout the US and Europe. Although combined modality data are limited for the use of ECP with radiation, one study has demonstrated disease free survival (DFS) and cause specific survival (CSS) advantage (after adjusting for B1 status and stage) for patients with erythrodermic mycosis fungoides who received a combination of ECP and total skin electron beam therapy (TSEBT) compared to TSBET without ECP. In a subset of these patients, persistent complete remissions have resulted from the therapy, suggesting that powerful and clinically relevant cytotoxic anti-tumor immune responses had been initiated. ECP has been distinguished from other forms of anti-cancer immunotherapy by both its efficacy and safety, but its evolution has been limited by the mystery of its mechanism. Recently, the key cellular components of ECP's efficacy, namely the simultaneous induction of apoptosis of malignant T cells and monocyte-to-dendritic cell (DC) conversion, have been recognized. Repetitive cycles of leukocyte adherence to and dissociation from the plastic (i.e. acrylic) faces of the ECP flow system device lead to the synchronous differentiation, within a single day, of processed monocytes into an extraordinarily large number (250 million) of immature DCs capable of internalizing apoptotic malignant cells and processing the expressed tumor antigens. This engineered phenomenon may be a mimicking of the normal conversion of monocytes to DCs as they insinuate themselves between endothelial cells to enter interstitial spaces.

Recently, we have found that overnight co-incubation of the two populations of induced cells, prior to their re-infusion, allows for more efficient cell-to-cell contact and processing of the apoptotic malignant T cells by the newly formed DCs, thus providing a rich source of tumor-loaded DCs in which all available tumor antigens are likely processed without the need to chemically isolate them or know their identity. We have termed the resulting transfer of immunizing tumor antigens to DC capable of stimulating specific anti-cancer immune responses "Transimmunization."

By incubating a patient's treated cells overnight, rather than returning them within two hours of photopheresis, as has been standard, we are able to increase the yield of dendritic cells. Rather than expose these DCs to malignant cells in vitro (in the overnight culture) as occurs in the treatment of CTCL, we propose to intravenously return the DCs to the patient-after overnight incubation in an effort to drive dendritic cell maturation-while the patient is undergoing a course of radiation therapy for NSCLC. Radiation therapy induces a cellular death via several mechanisms-including Apoptosis. Since intravenous return of the ECP-induced DCs would first (via the right heart) passage through the lung microvasculature, it is theorized that the DCs may gain access to the tumor. Direct anti-tumor effects by the DCs, as well as uptake of tumor cells/fragments and subsequent inductions of an anti-tumor response are potential beneficial consequences of the treatment.

The treatment involves the extracorporeal exposure of leukapheresed leukocytes to ultraviolet A activated 8-methoxypsoralen, a molecule naturally occurring in small quantities in a variety of plant products, including lime and celery. When this biologically inert furocoumarin is transiently activated by ultraviolet A energy, it is temporarily transformed into an alkylating agent which binds to pyrimidine bases of DNA. Since a single 8-MOP molecule is bivalent, cross-links between sister strands of DNA are formed, inhibiting both mitosis and gene function. It is important to note that while tumor cells will not be present in this mix (as is the case in leukemic cutaneous T cell lymphoma), and therefore will not be induced via 8-MOP/UVA exposure to undergo apoptosis, normal peripheral T cells that will be 8-MOP/UVA-induced into the apoptotic pathway are considered critical to driving monocytes to DC differentiation.

KLH (depyrogenated, endotoxin-free; Calbiochem-Novabiochem Corp., San Diego, CA) will be added at a concentration of 10 mg/ml to the DC-rich leukocyte culture prior to overnight culture. The cells will be placed in a CO2 incubator at 37° C overnight. The incubator will be committed solely to this purpose; only that patient's cells will be in it overnight; and it will be locked. The following morning, the patient's cells will be washed (i.e. centrifuged, re-suspended in 250 ml normal saline, and then centrifugated a second time) prior to being re-suspended in 250 mL of normal saline for infusion. The cells will be returned to the patient by intravenous infusion.

Side effects for standard photopheresis have been extremely limited and have required cessation of photopheresis in less than 1% of subjects. These side effects have most commonly included transient hypotension, due to the transient depletion in intravascular volume, which has been reversible on reinfusion of the blood, occasional difficulty in cannulating the antecubital vein, fever for a few hours following infusion of treated cells and elevation of serum uric acid, correctable with oral allopurinol administration. The current Phase I trial of transimmunization in the management of advanced CTCL in 26 individuals has suggested improved potency over conventional photopheresis, while maintaining the same excellent safety profile. As with its antecedent photopheresis, remarkably few adverse reactions have been experienced with transimmunization, and none of the subjects in the Phase I trial experienced limiting toxicity or required cessation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer Stage IIIB. Previously treated with two prior chemotherapy regimens or refused chemotherapy, and able to receive definitive RT. (Patients will not receive chemotherapy during the study). Patients with malignant pleural effusion are not eligible.
* Stage IV with measurable disease in the lung and a medical indication for radiation therapy. (Patients will not receive chemotherapy during the study). These patients must have received and progressed on two prior chemotherapy regimens or have refused chemotherapy.
* Staging by CT scan of chest/abdomen and MRI of brain.
* Willing and able to undergo two (baseline and follow-up) bronchoscopy with BAL and bronchial biopsy for bronchoscopically visible tumor.
* No treatment for lung cancer (chemotherapy, radiation therapy, biomodifiers) for 4 weeks prior to entry.
* Stable or progressive disease.
* No concurrent infection.
* Able to tolerate fluid shifts related to photopheresis (removal of 250 cc of blood and subsequent reinfusion of 250 cc of blood over 1-2 hours).
* ECOG Performance Status < 2.
* At least 18 years of age.
* Adequate bone marrow reserve: hemoglobin > 11 g/dL; platelet count > 100,000 mm3; ANC > 1500/ mL.
* Life expectancy of greater than 3 months.
* Normal peripheral CD8 count.
* Not pregnant or nursing.
* PFTs demonstrating diffusion capacity ≥ 60%, FEV1 ≥ 60%, and vital capacity ≥ 60%.
* Radiotherapy would be offered as appropriate standard therapy outside of a study setting.

Exclusion Criteria:

* History of or active infection with human immunodeficiency virus (HIV), hepatitis B (by antigenemia), or hepatitis C.
* History of allergic reactions attributed to compounds of similar composition to 8-methoxypsoralen (oxsoralen, trisoralen).
* Significant cardiovascular disease (i.e. NYHA class 3 or higher congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias)
* Pregnant or nursing at time of study entry.
* Participation in an investigational drug trial within 30 days prior to screening.
* Suspected or confirmed poor compliance, mental instability, or prior or current alcohol or drug abuse deemed by the Investigator to be likely to affect their ability to sign the informed consent, or undergo study procedures.
* Presentation with, or a recent history (within 24 hours) of a fever ≥ 38.2°C or symptoms of significant local infection or systemic infection, including urinary tract infections - such patients will be deferred from enrollment at least until 48 hours after illness has resolved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to determine the safety of using a treatment called transimmunization in addition to standard therapy (radiation) in the treatment of lung cancer. | 1-2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Emil Bisaccia, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States